CLINICAL TRIAL: NCT04437602
Title: Added Value of Preoperative Contrast Enhanced Mammography (PROCEM) in Staging of Malignant Breast Lesions - a Prospective Randomized Multicenter Trial
Brief Title: Added Value of Preoperative Contrast Enhanced Mammography in Staging of Malignant Breast Lesions
Acronym: PROCEM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Halland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-02661
Record Dates: First submitted 2020-05-27; First posted 2020-06-18 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
Keywords: Contrast Enhanced Mammography; Preoperative staging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CEM (Experimental): Patients in experimental arm will go through additional preoperative staging with contrast enhanced mammography
  Interventions: Diagnostic Test: Contrast Enhanced Mammography (CEM)
- No CEM (No Intervention): Patients in No intervention arm will go through no additional preoperative imaging

INTERVENTIONS:
Diagnostic Test: Contrast Enhanced Mammography (CEM) — Additional CEM in preoperative staging
  Arms: CEM

SUMMARY:
Patients diagnosed with breast cancer after routine assessment with digital mammography and ultrasound and scheduled for primary surgery are included in the trial. The patients are randomized 1:1 to go through additional contrast enhanced mammography (CEM) or no further imaging preoperatively. Primary endpoint is rate of patients with change of treatment: a) mastectomy instead of partial mastectomy due larger unifocal or multifocal extent, b) partial mastectomy instead of mastectomy due to improved demarcation of the tumour area, c) bilateral surgery instead of unilateral due to findings of contralateral cancer, d) neoadjuvant therapy instead of primary surgery due to more advanced disease. Rate of reoperation and rate of avoidable mastectomies are secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Planned primary surgery for suspicious or verified breast malignancy Age of 18 years and above Signed informed consent

Exclusion Criteria:

* Planned neoadjuvant therapy On-going pregnancy Iodinated contrast agent allergy Renal failure (abnormal S-creatinine) Untreated thyreotoxicosis Severe heart failure Myastenia gravis Breast implant Local recurrence as index lesion Inability to understand and comprehend oral and written information of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer is very uncommon among men.
Enrollment: 441 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with change of primary treatment due to findings at additional CEM | Within two months after diagnosis of breast cancer
  Mastectomy instead of partial mastectomy due to findings of multifocal disease, mastectomy instead of partial mastectomy due to larger unifocal extent, partial mastectomy instead of mastectomy due to improved demarcation of tumour area, bilateral surgery due to findings of contralateral cancer, primary neoadjuvant treatment instead of primary surgery due to more advanced disease

SECONDARY OUTCOMES:
Rate of reoperations | Within three months after diagnosis of breast cancer
  Number of reoperations due to inadequate margins
Rate of avoidable mastectomies | Within three months after diagnosis of breast cancer
  Patients operated with mastectomy where histopathology shows extent less than 3 cm

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Ahsberg, PhD, Principal Investigator — Region Halland
Locations (3):
- Sweden (3):
  - Halland Hospital Halmstad, Halmstad
  - Helsingborg Hospital, Helsingborg
  - Central Hospital Kristianstad, Kristianstad

IPD SHARING:
Plan to Share IPD: No
No plan

REFERENCES:
- [Background] Ahsberg K, Gardfjell A, Nimeus E, Ryden L, Zackrisson S. The PROCEM study protocol: Added value of preoperative contrast-enhanced mammography in staging of malignant breast lesions - a prospective randomized multicenter study. BMC Cancer. 2021 Oct 18;21(1):1115. doi: 10.1186/s12885-021-08832-2. PMID 34663236
- [Result] Ahsberg K, Gardfjell A, Nimeus E, Rasmussen R, Behmer C, Zackrisson S, Ryden L. Added value of contrast-enhanced mammography (CEM) in staging of malignant breast lesions-a feasibility study. World J Surg Oncol. 2020 May 21;18(1):100. doi: 10.1186/s12957-020-01865-0. PMID 32438917